CLINICAL TRIAL: NCT01151020
Title: Zenith® TX2® Low Profile TAA Endovascular Graft Clinical Study
Brief Title: TX2® Low Profile TAA Endovascular Graft
Acronym: TX2® LP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cook Research Incorporated (Industry)
Responsible Party: Sponsor
Organization: Cook Group Incorporated (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-001; NCT00923754 (obsolete NCT alias)
Expanded Access: NCT02471781 (Approved for marketing)
Record Dates: First submitted 2010-06-22; First posted 2010-06-25 (Estimated); Results first posted 2016-02-29 (Estimated); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Aortic Aneurysm; Penetrating Ulcer; Vascular Disease
Keywords: Aortic Aneurysm; Aneurysm; Vascular Prosthesis; Vascular Disease; Blood Vessel Prosthesis Implantation
MeSH Terms: conditions — Aortic Aneurysm; Penetrating Atherosclerotic Ulcer; Vascular Diseases; Aneurysm | interventions — Endovascular Aneurysm Repair

ARMS (1):
- Arm 1 (Experimental): Zenith® TX2® Low Profile TAA Endovascular Graft (Thoracic Aortic Aneurysm)
  Interventions: Device: Zenith® TX2® Low Profile TAA Endovascular Graft

INTERVENTIONS:
Device: Zenith® TX2® Low Profile TAA Endovascular Graft — Endovascular treatment of patients with aneurysms/ulcers of the descending thoracic aorta having morphology suitable for endovascular repair
  Other Names: Zenith Alpha Thoracic™ Endovascular Graft; TEVAR

SUMMARY:
The Zenith® TX2® Low Profile TAA Endovascular Graft study is a clinical trial approved by US FDA to evaluate the safety and effectiveness of the Zenith® TX2® Low Profile TAA Endovascular Graft indicated for the treatment of patients with aneurysms/ulcers of the descending thoracic aorta having vessel structure suitable for repair.

ELIGIBILITY:
Inclusion Criteria:

* Descending thoracic aneurysm with diameter ≥ 5.0 cm
* Descending thoracic aneurysm with a history of growth ≥ 0.5 cm per year
* Descending thoracic degenerative or atherosclerotic ulcer ≥ 10 mm in depth and 20 mm in diameter

Exclusion Criteria:

* Less than 18 years of age
* Life expectancy less than 2 years
* Pregnant or breastfeeding or planning on becoming pregnant within 60 months
* Unwilling to comply with the follow-up schedule
* Inability or refusal to give informed consent
* Less than 30 days beyond primary endpoint for other investigative drug or device study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2010-03; Primary Completion 2014-01 (Actual); Study Completion 2018-05-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karl Illig, MD, Principal Investigator — University of South Florida
Locations (33):
- United States (22):
  - Kaiser Permanente, San Francisco, California
  - Washington Hospital Center, Washington D.C., District of Columbia
  - University of South Florida, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Methodist Hospital of Indiana, Indianapolis, Indiana
  - Indiana Heart Hospital, Indianapolis, Indiana
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Cooper University Hospital, Camden, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - New York University Hospital, New York, New York
  - Mount Sinai Hospital, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Tennessee Baptist Memorial Hospital, Memphis, Tennessee
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Harborview Medical Center, Seattle, Washington
- Germany (5):
  - Hannover Medical School, Hanover
  - St. Franziskus Hospital, Münster
  - Klinikum Nürnberg Sud, Nuremberg
  - Uniklinik Regensburg, Regensburg
  - University Hospital Rostock, Rostock
- Hospital San Raffaele, Milan, Italy
- Japan (3):
  - Morinomiya Hospital, Osaka
  - Jikei University School of Medicine, Tokyo
  - Keio University Hospital, Tokyo
- Malmö University Hospital, Malmo, Sweden
- St.George's Hospital, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Zenith® TX2® Low Profile TAA Endovascular Graft
Started | 110
30-day | 110
Completed | 56
Not Completed | 54
Not completed — Death | 25
Not completed — Conversion to open repair | 1
Not completed — Lost to Follow-up | 4
Not completed — Withdrawal by Subject | 22
Not completed — Patients did not receive the device | 2

BASELINE CHARACTERISTICS:
Arm/Group | Zenith® TX2® Low Profile TAA Endovascular Graft
Number analyzed (Participants) | 110
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.2 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46
  Male | 64

OUTCOME MEASURES:

1. Primary Outcome: Patients With Major Adverse Events (MAE)
Description: Major adverse event is defined as:
  All-cause death; Q-wave MI; cardiac event involving arrest, resuscitation, or balloon pump; ventilation > 72 hours or re-intubation; pulmonary event requiring tracheostomy or chest tube; renal failure requiring permanent dialysis, hemofiltration, or kidney transplant in a patient with a normal pre-procedure serum creatinine level; bowel resection; stroke; paralysis; amputation involving more than toes; aneurysm or vessel leak requiring re-operation; deep vein thrombosis requiring surgical or lytic therapy; pulmonary embolism involving hemodynamic instability or surgery; coagulopathy requiring surgery; or wound complication requiring return to the operating room.
Time Frame: 30 days
Population: 1 patient had a stroke and required ventilation >72 hours/reintubation.
Measure: Number; unit: participants
Arm/Group | Zenith® TX2® Low Profile TAA Endovascular Graft
Number analyzed (Participants) | 110
participants
  Stroke | 2
  Ventilation >72 hours/reintubation | 3
Statistical Analysis 1: Comparison: Zenith® TX2® Low Profile TAA Endovascular Graft; Null hypothesis: The 30-day freedom from MAE for patients treated with the Zenith® TX2® Low Profile TAA Endovascular Graft does not meet the performance goal of 80.6%; Test type: Superiority or Other; p < 0.001, Exact binomial test; Free from major adverse event rate (%) = 96.4, 95% CI 2-sided [91 to 99]

2. Primary Outcome: Patients With Device Failures
Description: Device failure is defined as: Technical failure (inability to access or deploy the Zenith® TX2® Low Profile TAA Endovascular Graft or loss of patency at the time of deployment completion), or any of the following: type I or type III endoleaks requiring re-intervention, aneurysm rupture or conversion to open surgical repair, aneurysm enlargement greater than 0.5 cm.
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | Zenith® TX2® Low Profile TAA Endovascular Graft
Number analyzed (Participants) | 110
participants
  Did not receive the device (technical failures) | 2
  Aneurysm growth>5 mm | 2
  Aneurysm growth>5 mm and conversion to open repair | 1
  Endoleak requiring secondary intervention | 3
Statistical Analysis 1: Comparison: Zenith® TX2® Low Profile TAA Endovascular Graft; Null Hypothesis: The 12-month device success for patients treated with the Zenith® TX2® Low Profile TAA Endovascular Graft does not meet the performance goal of 80.7%; Test type: Superiority or Other; p < 0.001, Exact binomial test; Device success rate (%) = 92.7, 95% CI 2-sided [86.2 to 96.8]

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | Zenith® TX2® Low Profile TAA Endovascular Graft
All-Cause Mortality (participants affected / at risk) | 25/110
Serious Adverse Events (participants affected / at risk) | 86/110
Other Adverse Events (participants affected / at risk) | 0/110
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zenith® TX2® Low Profile TAA Endovascular Graft (N=110)
coagulopathy (Blood and lymphatic system disorders) | 1 (1)
Arrhythmia (Cardiac disorders) | 1 (1)
thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
angina pectoris (Cardiac disorders) | 1 (2)
cardiac arrest (Cardiac disorders) | 1 (1)
cardiac failure congestive (Cardiac disorders) | 5 (5)
myocardial infarction (Cardiac disorders) | 6 (7)
myocardial ischaemia (Cardiac disorders) | 1 (1)
ventricular tachycardai (Cardiac disorders) | 1 (1)
Intestinal Ischaemia (Gastrointestinal disorders) | 4 (4)
aorto-oesophageal fistula (Gastrointestinal disorders) | 1 (1)
dysphagia (Gastrointestinal disorders) | 1 (1)
ileus (Gastrointestinal disorders) | 1 (1)
inguinal hernia (Gastrointestinal disorders) | 2 (2)
pneumoperitoneum (Gastrointestinal disorders) | 1 (1)
Vascular injury (Injury, poisoning and procedural complications) | 1 (1)
brain contusion (Injury, poisoning and procedural complications) | 1 (1)
femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1)
foreign body (Injury, poisoning and procedural complications) | 1 (1)
incisional hernia (Injury, poisoning and procedural complications) | 1 (1)
injury (Injury, poisoning and procedural complications) | 1 (1)
patella fracture (Injury, poisoning and procedural complications) | 1 (1)
spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1)
subdural hematoma (Injury, poisoning and procedural complications) | 1 (1)
compartment syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
spinal ligament ossification (Musculoskeletal and connective tissue disorders) | 1 (2)
spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Gastric cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
blindness unilateral (Eye disorders) | 1 (1)
cataract (Eye disorders) | 1 (1)
abdominal pain lower (Gastrointestinal disorders) | 1 (1)
gastrointestinal haemorrhage (Gastrointestinal disorders) | 5 (5)
intestinal obstruction (Gastrointestinal disorders) | 1 (1)
oesophageal dysplasia (Gastrointestinal disorders) | 1 (1)
pelvic floor dysfunction (Gastrointestinal disorders) | 1 (1)
small intestinal obstruction (Gastrointestinal disorders) | 3 (3)
chest pain (General disorders) | 2 (2)
multiple organ dysfunction syndrome (General disorders) | 2 (2)
stent-graft endoleak (General disorders) | 7 (7)
cholecystitis acute (Hepatobiliary disorders) | 1 (1)
anaphylactic reaction (Immune system disorders) | 1 (1)
contrast media allergy (Immune system disorders) | 1 (1)
abdominal wall abscess (Infections and infestations) | 1 (1)
abdominal wall infection (Infections and infestations) | 1 (1)
arthritis bacterial (Infections and infestations) | 1 (1)
diverticulitis (Infections and infestations) | 1 (1)
diverticulitis intestinal perforated (Infections and infestations) | 1 (1)
gastroenteritis (Infections and infestations) | 1 (1)
gastrointestinal infection (Infections and infestations) | 5 (5)
infection (Infections and infestations) | 1 (1)
influenza (Infections and infestations) | 1 (1)
pneumonia (Infections and infestations) | 12 (13)
sepsis (Infections and infestations) | 2 (2)
urinary tract infection (Infections and infestations) | 2 (2)
fall (Injury, poisoning and procedural complications) | 3 (3)
hip fracture (Injury, poisoning and procedural complications) | 1 (1)
post laminectomy syndrome (Injury, poisoning and procedural complications) | 1 (1)
pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1)
respiratory fume inhalation disorder (Injury, poisoning and procedural complications) | 1 (1)
spinal column injury (Injury, poisoning and procedural complications) | 1 (1)
blood creatinine increased (Investigations) | 3 (3)
gout (Metabolism and nutrition disorders) | 1 (1)
malnutrition (Metabolism and nutrition disorders) | 1 (1)
arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1)
lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Generalized tonic-clonic seizure (Nervous system disorders) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1)
aphasia (Nervous system disorders) | 1 (1)
carotid artery stenosis (Nervous system disorders) | 1 (1)
cerebrovascular accident (Nervous system disorders) | 8 (8)
paraparesis (Nervous system disorders) | 1 (1)
parkinsonism (Nervous system disorders) | 1 (1)
syncope (Nervous system disorders) | 2 (2)
device electrical finding (Product Issues) | 1 (1)
delirium (Psychiatric disorders) | 1 (1)
Nephropathy toxic (Renal and urinary disorders) | 1 (1)
calculus urinary (Renal and urinary disorders) | 1 (1)
chronic kidney disease (Renal and urinary disorders) | 1 (1)
renal failure (Renal and urinary disorders) | 6 (7)
urinary incontinence (Renal and urinary disorders) | 1 (1)
prostatitis (Reproductive system and breast disorders) | 1 (1)
acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
aorto-bronchial fistula (Respiratory, thoracic and mediastinal disorders) | 1 (1)
bronchial secretion retention (Respiratory, thoracic and mediastinal disorders) | 1 (1)
chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2)
haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
pulmonary haematoma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Soft tissue excision (Surgical and medical procedures) | 1 (1)
craniotomy (Surgical and medical procedures) | 1 (1)
percutaneous coronary intervention (Surgical and medical procedures) | 1 (1)
Aneurysm (Vascular disorders) | 14 (15)
aortic aneurysm (Vascular disorders) | 2 (2)
embolism (Vascular disorders) | 3 (3)
haematoma (Vascular disorders) | 1 (1)
haemmorrhage (Vascular disorders) | 1 (1)
hypertension (Vascular disorders) | 1 (1)
hypotension (Vascular disorders) | 1 (1)
iliac artery occlusion (Vascular disorders) | 1 (1)
iliac artery stenosis (Vascular disorders) | 2 (2)
ischaemia (Vascular disorders) | 1 (1)
peripheral arterial occlusive disease (Vascular disorders) | 1 (1)
peripheral artery occlusion (Vascular disorders) | 1 (1)
vascular dissection (Vascular disorders) | 3 (3)
vascular rupture (Vascular disorders) | 3 (3)
ATRIAL FIBRILLATION (Cardiac disorders) | 1 (1)
CARDIAC FAILURE (Cardiac disorders) | 1 (3)
CORONARY ARTERY STENOSIS (Cardiac disorders) | 1 (1)
RETROPERITONEAL HAEMATOMA (Gastrointestinal disorders) | 1 (1)
DEATH (General disorders) | 2 (2)
VASCULAR STENT THROMBOSIS (General disorders) | 1 (1)
CHOLANGITIS (Hepatobiliary disorders) | 1 (1)
CHOLELITHIASIS (Hepatobiliary disorders) | 1 (1)
OSTEOMYELITIS (Infections and infestations) | 1 (1)
HERPES ZOSTER (Infections and infestations) | 1 (1)
ABSCESS LIMB (Infections and infestations) | 1 (1)
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
POST PROCEDURAL HAEMMORRHAGE (Injury, poisoning and procedural complications) | 1 (1)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
BONE METABOLISM DISORDER (Musculoskeletal and connective tissue disorders) | 1 (1)
MUSCLE RUPTURE (Musculoskeletal and connective tissue disorders) | 1 (1)
POLYMYALGIA RHEUMATICA (Musculoskeletal and connective tissue disorders) | 1 (1)
URETHRAL STENOSIS (Renal and urinary disorders) | 1 (1)
URINARY RETENTION (Renal and urinary disorders) | 2 (2)
LUNG OPACITY (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PULMONARY CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1 (1)
DECUBITUS ULCER (Skin and subcutaneous tissue disorders) | 1 (1)
STASIS DERMATITIS (Skin and subcutaneous tissue disorders) | 1 (1)
MEDICAL DEVICE REMOVAL (Surgical and medical procedures) | 1 (1)
RENAL DISORDER PROPHYLAXIS (Surgical and medical procedures) | 2 (3)
STENT PLACEMENT (Surgical and medical procedures) | 1 (1)
ABDOMINAL ADHESIONS (Gastrointestinal disorders) | 1 (1)
PAPILLA OF VATER STENOSIS (Gastrointestinal disorders) | 1 (1)
MULTIPLE FRACTURES (Injury, poisoning and procedural complications) | 1 (1)
BURSITIS (Injury, poisoning and procedural complications) | 1 (1)
MENTAL STATUS CHANGES (Psychiatric disorders) | 1 (1)
DEPENDENCE ON VENTILATOR (Respiratory, thoracic and mediastinal disorders) | 1 (1)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days